CLINICAL TRIAL: NCT01755208
Title: Light-Scattering Spectroscopy for the Detection of Stage II-III Breast Cancer: A Pilot Study
Brief Title: Light-Scattering Spectroscopy for Detection of Breast Cancer
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Insufficient Accrual
Sponsor: University of Southern California (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 1B-12-6; NCI-2012-02769 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2012-12-18; First posted 2012-12-24 (Estimated); Last update posted 2021-11-19 (Actual); Status verified 2021-11

CONDITIONS: Healthy, no Evidence of Disease; Stage II Breast Cancer; Stage IIIA Breast Cancer; Stage IIIB Breast Cancer; Stage IIIC Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Diagnostic (light-scattering spectroscopy) (Experimental): Patients undergo light-scattering spectroscopy of the breast in addition to standard of care as it relates to screening for breast cancer or treatment of breast cancer.
  Interventions: Procedure: light-scattering spectroscopy

INTERVENTIONS:
Procedure: light-scattering spectroscopy — Undergo light-scattering spectroscopy

SUMMARY:
This pilot clinical trial studies light-scattering spectroscopy in finding disease in patients with stage II-III breast cancer. Diagnostic procedures, such as light-scattering spectroscopy, may help find and diagnose breast cancer

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES: I. To evaluate whether light-scattering spectroscopy can reliably distinguish between two subject groups: those with clinical stage II or stage III breast cancer and those without breast cancer.

OUTLINE: Patients undergo light-scattering spectroscopy of the breast in addition to standard of care as it relates to screening for breast cancer or treatment of breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Participants who are breast cancer free (mammogram "negative" within 1 month of testing) with the absence of clinical suspicion of breast cancer on physical exam or with clinical stage II or stage III breast cancer. PLEASE NOTE: Recruitment for this study is only limited to patients who are scheduled for a mammogram at USC. There is no compensation to participants.
* Provision of informed consent prior to any study-related procedures

Exclusion Criteria:

* Females with tattoos on either or both breasts
* Females with nipple piercings on either or both breasts
* Females with skin piercings (aka microdermal anchor surface or microdermal piercings) in either or both breasts
* Females unable to provide informed consent
* Females s/p treatment for breast cancer

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2012-11-21 (Actual); Primary Completion 2020-11-19 (Actual); Study Completion 2020-11-19 (Actual)

PRIMARY OUTCOMES:
Accurate classifications of women with or without breast cancer | Up to 1 year
  Exact binomial probabilities will be used.
Utility of optical markers in distinguishing cancer involved breasts from normal breasts | Up to 1 year
  Multivariate analyses will be used.

CONTACTS AND LOCATIONS:
Overall Officials: Jacques Van Dam, Principal Investigator — University of Southern California
Locations (1):
- USC Norris Comprehensive Cancer Center, Los Angeles, California, United States